CLINICAL TRIAL: NCT03079076
Title: Ultrasound Guided Modified Thoracolumbar Interfascial Plane Block for Spinal Surgery: A New Approach
Brief Title: Ultrasound Guided Modified Thoracolumbar Interfascial Plane Block for Spinal Surgery
Acronym: TLIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, MD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUTF ANESTHESIA4
Record Dates: First submitted 2017-03-06; First posted 2017-03-14 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Pain, Postoperative; Spine Disease
Keywords: Postoperative Analgesia; Ultrasound guided thoracolumbar interfascial plane block
MeSH Terms: conditions — Pain, Postoperative; Spinal Diseases | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thoracolumbar interfascial plane block (Active Comparator): Bilateral ultrasound guided thoracolumbar interfascial plane block with 20 ml %0,25 bupivacaine
  Interventions: Drug: Bupivacaine
- sham block (Placebo Comparator): Bilateral ultrasound guided sham block with 2 ml saline subcutaneously
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — 20 ml %0,25 bupivacaine bilaterally
  Other Names: ultrasound guided thoracolumbar interfascial plane block
  Arms: thoracolumbar interfascial plane block
Drug: Saline — 2 ml saline subcutaneously bilaterally
  Other Names: ultrasound guided sham block
  Arms: sham block

SUMMARY:
Ultrasound guided thoracolumbar interfascial plane (TLIP) block was first described in 2015 by Hand et al. TLIP block involves injection of local anesthetics between multifidus and longissimus muscles at the third lumbar vertebra level and can block the dorsal rami of thoracolumbar nerves. In new approach differently, the investigators made the injection between longissimus and iliocostalis muscles with a 15 degree angle from medial to lateral.

The aim of this study is to determine effectiveness of ultrasound guided thoracolumbar interfascial plane (TLIP) block in patients undergoing spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients undergoing spinal surgery

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | First 24 hours total opioid consumption
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | postoperative first hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at first hour postoperatively
Visual analog pain score | postoperative second hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at second hour postoperatively.
Visual analog pain score | postoperative 4th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 4th hour postoperatively
Visual analog pain score | postoperative 8th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 8th hour postoperatively
Visual analog pain score | postoperative 12th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 12th hour postoperatively.
Visual analog pain score | postoperative 24th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 24th hour postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600
- [Background] Ahiskalioglu A, Alici HA, Selvitopi K, Yayik AM. Ultrasonography-guided modified thoracolumbar interfascial plane block: a new approach. Can J Anaesth. 2017 Jul;64(7):775-776. doi: 10.1007/s12630-017-0851-y. Epub 2017 Feb 27. No abstract available. PMID 28243853
- [Background] Ueshima H, Oku K, Otake H. Ultrasound-guided thoracolumbar interfascial plane block: a cadaveric study of the spread of injectate. J Clin Anesth. 2016 Nov;34:259-60. doi: 10.1016/j.jclinane.2016.04.060. Epub 2016 May 13. No abstract available. PMID 27687388 (Retraction: PMID 35393195 J Clin Anesth. 2022 Aug;79:110771)